CLINICAL TRIAL: NCT01968291
Title: The Impact of Teach-back on Comprehension of Discharge Instructions Among Emergency Patients With Limited Health Literacy: A Randomized, Controlled Study
Brief Title: Use of Teach Back to Improve Comprehension of Discharge Instructions for Emergency Patients With Limited Health Literacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Richard Griffey, Associate Professor, Emergency Medicine, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 201206011
Record Dates: First submitted 2013-10-10; First posted 2013-10-24 (Estimated); Last update posted 2013-10-24 (Estimated); Status verified 2013-10

CONDITIONS: Conditions Influencing Health Status
Keywords: Health Literacy; Teach-back; Emergency
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Teach-back (Experimental): Patients are prompted to state back in their own words their comprehension of the information given to them at discharge.
  Interventions: Behavioral: Teach-back
- Standard Discharge Instructions (No Intervention): Patient receives usual discharge instructions as administered by the nurse assigned to the patient.

INTERVENTIONS:
Behavioral: Teach-back — Patients are asked to repeat back in their own words their understanding of the discharge information that was provided to them.
  Arms: Teach-back

SUMMARY:
The purpose of this study was to determine whether use of teach-back discharge instructions improve patient satisfaction and patients' self-reported and objective comprehension of discharge instructions in the emergency department when compared to standard discharge instructions.

ELIGIBILITY:
Inclusion Criteria:

* patients being discharged from the emergency department
* A score of 6 or less on the Rapid Estimate of Adult Literacy in Medicine, Revised (consistent with Limited Health Literacy)

Exclusion Criteria:

* aphasia,
* non-English speaking,
* mental handicap,
* psychiatric chief complaint,
* too high acuity per physician,
* insurmountable communication barrier,
* evaluations for sexual assault,
* clinical intoxication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2012-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Objective comprehension | Questions evaluating comprehension were administered during the discharge interview immediately following discharge from the ED at the index visit (Day 1).
  Concordance between audio taped comprehension compared to review of medical record using 5 level scale of concordance

SECONDARY OUTCOMES:
self-reported comprehension | Questions evaluating self-reported comprehension were administered during the discharge interview immediately following discharge from the ED at the index visit (Day 1).
  self reported comprehension of discharge instructions for the following areas: emergency department (ED) course (Tests and treatment); Post-ED care (medication instructions; home instructions; follow-up instructions); Return instructions.

OTHER OUTCOMES:
patient satisfaction | Questions evaluating satisfaction were administered during the discharge interview immediately following discharge from the ED at the index visit (Day 1).
  Patient satisfaction as measured by 4 questions modified from the Consumer Assessment of Health Providers & Systems (CAHPS) Clinician & Group Surveys

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Griffey, MD, MPH, Principal Investigator — Washington University School of Medicine; Kim A Kaphingst, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Barnes-Jewish Hospital Emergency Department, St Louis, Missouri, United States